CLINICAL TRIAL: NCT04710875
Title: The Role of Lactate in Lipolysis and Catabolism in Humans
Acronym: LILACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1-10-72.180-20
Record Dates: First submitted 2020-12-01; First posted 2021-01-15 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2020-09

CONDITIONS: Hyperlactatemia; Healthy; Lactate
Keywords: Lipolysis; Catabolism; Glucose metabolism; Aminoacid metabolisme
MeSH Terms: conditions — Hyperlactatemia | interventions — Sodium Lactate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Na-lactate (Active Comparator): Iv infusion of sodium D/L lactate
  Interventions: Drug: Na-lactate
- Sodium chloride (Placebo Comparator): Iv infusion of Sodium chloride
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Na-lactate — intravenous
  Other Names: Sodium lactate
  Arms: Na-lactate
Drug: Sodium chloride — Intravenous
  Other Names: NaCl
  Arms: Sodium chloride

SUMMARY:
Lactate may have anti-lipolytic effects when plasma concentrations of lactate reach levels similar to those seen during high intensity exercise.

This study aims to investigate how lactate concentrations similar to those achieved during high intensity exercise affects lipolysis in humans. In addition to this, to investigate how increased lactate concentrations affects glucose- and amino acid metabolism.

8 healthy males will be included. Study participants will undergo two separate investigation days that will be identical except for the interventions:

1. Intravenous sodium D/L-lactate
2. Intravenous sodium chloride.

The study consists of a 3-hour basal period followed by a 3-hour hyperinsulinemic euglycemic clamp. During the study we will:

* Estimate insulin sensitivity during the hyperinsulinemic euglycemic clamp (M value)
* Use tracer kinetics to estimate lipid-, glucose and amino acid metabolism using [9,10-3H]-palmitate, [3-3H]-glucose, [15N]-phenylalanine, [15N]-tyrosine, [2H4]-tyrosine and [13C]-Urea.
* Do muscle- and adipose tissue biopsies for analyses of signaling pathways involved in regulation of lipid-, glucose and amino acid metabolism.
* Do blood samples of relevant hormones, metabolites and cytokines.
* Use indirect calorimetry to estimate study participants' resting energy expenditure and respiratory quotient during the basal period.
* Estimate cardiac ejection fraction by echocardiography and measure blood pressure during both the basal- and clamp period.

ELIGIBILITY:
Inclusion Criteria:

* male
* >18 years of age
* BMI >19 and below 30
* Written and verbal consent to participation

Exclusion Criteria:

* Chronic illness
* daily use of medicine
* affected blood samples at screening, as assessed by the PI
* does not speak and understand Danish
* Assessed unsuitable by PI.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Acute Metabolic effects of Na-lactate compared with NaCl on lipolysis | 2 hours (1 hour basal period, 1 hour clamp)
  Change in [9,10-3H]-palmitate tracer flux

SECONDARY OUTCOMES:
Acute Metabolic effects of Na-lactate compared with NaCl on glucose metabolism | 6 hours (3 hours basal period, 3 hours clamp)
  Change in glucose metabolism quantified with [3-3H]-glucose tracer
Insulin sensitivity | 3 hours.
  Hyperinsulinaemic euglycaemic clamp with 0.6mU/kg/min insulin and 20% glucose to calculate M value. Difference between interventions.
Acute metabolic effects of Na-lactate compared with NaCl on aminoacid metabolism | 6 hours
  Change in aminoacid metabolism quantified with [15N]-phenylalanine, [15N]tyrosine, [2H4]tyrosine and [13C]-Urea tracers.
Indirect calorimetry during clamp | 20 minutes
  Change in estimation of resting energy expenditure during clamp. Difference between interventions.
Indirect calorimetry during basal conditions | 20 minutes
  Change in estimation of respiratory quotient during basal period. Difference between interventions.
Echocardiography | 15 minutes
  Change in cardiac ejection fraction during basal period. Difference between interventions.
Echocardiography | 15 minutes
  Change in cardiac ejection fraction during clamp period. Difference between interventions.
blood pressure | 2 x 10 min
  blood pressure (systolic and diastolic) during basal- and clamp
Blood samples - Insulin | 6 hours.
  Insulin concentrations. Difference between interventions.
Blood samples - c-peptid | 6 hours.
  c-peptid concentrations. Difference between interventions.
Blood samples - glucagon | 6 hours.
  glucagon concentrations. Difference between interventions.
Blood samples - cortisol | 6 hours.
  cortisol concentrations. Difference between interventions.
Blood samples - Ghrelin | 6 hours.
  Ghrelin concentrations. Difference between interventions.
Blood samples - GDF-15 | 6 hours.
  GDF-15 concentrations. Difference between interventions.
Blood samples - free fatte acids | 6 hours.
  Free fatte acids concentrations. Difference between interventions.
Blood samples - glucose | 6 hours.
  glucose concentrations. Difference between interventions.
Blood samples - lactate | 6 hours.
  lactate concentrations. Difference between interventions.
Changes in signaling in muscle tissue between interventions | After 3 and 5 hours of intervention
  Western blot examinations of muscle tissue biopsies
Changes in signaling in adipose tissue between interventions | After 3 and 5 hours of intervention
  Western blot examinations of adipose tissue biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Niels Møller, Prof, MD, DMSc, Study Director — Medical/Steno Aarhus research laboratory, Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Medical/Steno Aarhus research laboratory, Aarhus, Central Region Denmark
  - Aarhus University Hospital, Aarhus N

REFERENCES:
- [Derived] Berg-Hansen K, Gopalasingam N, Pedersen MGB, Nyvad JT, Rittig N, Sondergaard E, Wiggers H, Moller N, Nielsen R. Cardiovascular effects of lactate in healthy adults. Crit Care. 2025 Jan 17;29(1):30. doi: 10.1186/s13054-025-05259-0. PMID 39825426